CLINICAL TRIAL: NCT03503578
Title: Electroencephalogram Studies of Induction and Recovery From Sevoflurane-Induced General Anesthesia
Brief Title: EEG Studies of Sevoflurane-Induced General Anesthesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Oluwaseun Johnson-Akeju, MD, MMSc, Associate Professor of Anaesthesia, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 2014P000111
Record Dates: First submitted 2018-04-05; First posted 2018-04-20 (Actual); Results first posted 2019-10-24 (Actual); Last update posted 2019-10-24 (Actual); Status verified 2019-10

CONDITIONS: Anesthesia
MeSH Terms: interventions — Sevoflurane; Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- EEG Dynamics (Experimental): EEG data will be collected on patients receiving sevoflurane, and sevoflurane and ketamine together.
  Interventions: Drug: Sevoflurane; Drug: Ketamine

INTERVENTIONS:
Drug: Sevoflurane — Subjects will received sevoflurane for approximately 60 minutes.
Drug: Ketamine — Subjects will received sevoflurane and ketamine for approximately 60 minutes.

SUMMARY:
The investigators are performing this research study to find out how and where the anesthetic drugs sevoflurane and ketamine act in the brain. Sevoflurane and ketamine are anesthetics (a drug or agent used to decrease or eliminate the feeling of pain by causing unconsciousness). The investigators will study the brain using a machine that records the brain's electrical activity, called an electroencephalogram (EEG).

DETAILED DESCRIPTION:
During this research study, participants will receive sevoflurane, and sevoflurane and ketamine together, at a high enough dose to induce general anesthesia (make study participants "fall asleep"). During one visit participants will receive only sevoflurane; during another visit participants will be given both sevoflurane and ketamine together. The investigators will record EEG the entire time. The investigators will also ask some questions related to pain and cognitive function.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 50
* Normal body weight and habitus, BMI ≤ 30
* Non-smoker
* American Society of Anesthesiologists (ASA) physical status classification P1

Exclusion Criteria:

* Chronic health conditions

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-08-01 (Actual); Study Completion 2018-08-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | EEG Dynamics
Started | 12
Completed | 12
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | EEG Dynamics
Number analyzed (Participants) | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 25 (4.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 11
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 8
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Frequencies At Which Changes in Alpha, Theta, and Slow-Delta Wave Power Were Observed From Baseline During Sevoflurane-induced General Anesthesia
Description: Changes in power from baseline at various EEG spectral frequencies were assessed at sevoflurane-induced loss of responsiveness. EEGs of 12 patients were analyzed to determine changes in various EEG spectral frequencies (alpha, theta, delta, etc.) from baseline. The outcome measure reflects the associated frequency (Hz) at which changes were found under sevoflurane-induced general anesthesia. These frequency values are a representation of the findings for all 12 participants.
Time Frame: Approximately 60 minutes
Measure: Number; unit: Hz
Groups:
- EEG Dynamics: EEG data will be collected on patients receiving sevoflurane anesthesia.
Arm/Group | EEG Dynamics
Number analyzed (Participants) | 12
Hz
  Alpha | 10
  Theta | 5
  Slow-Delta | 1

ADVERSE EVENTS:
Time Frame: From initiation of anesthesia during the first study visit to completion of the second study visit. Study visits typically occurred less than 1 week apart.
Description: Adverse events and other events were determined by regular investigator assessment and self-reporting.
Arm/Group | EEG Dynamics
All-Cause Mortality (participants affected / at risk) | 0/12
Serious Adverse Events (participants affected / at risk) | 0/12
Other Adverse Events (participants affected / at risk) | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-24): https://cdn.clinicaltrials.gov/large-docs/78/NCT03503578/Prot_SAP_000.pdf